CLINICAL TRIAL: NCT02068339
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of Oltipraz for Liver Fat Reduction in Patients With Non-Alcoholic Fatty Liver Disease Except for Liver Cirrhosis
Brief Title: Efficacy and Safety of Oltipraz for Liver Fat Reduction in Patients With Non-Alcoholic Fatty Liver Disease Except for Liver Cirrhosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PharmaKing (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PMK-N01GI1_Phase 3
Record Dates: First submitted 2014-02-19; First posted 2014-02-21 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Non-alcholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo Comparator / Tid (total 0mg)
  Interventions: Drug: Placebo
- Oltipraz 1 (Experimental): Total 90mg, by mouth, tid
  Interventions: Drug: Oltipraz 1 (90mg)
- Oltipraz 2 (Experimental): Total 120mg, by mouth, tid
  Interventions: Drug: Oltipraz 2 (120mg)

INTERVENTIONS:
Drug: Oltipraz 1 (90mg)
  Arms: Oltipraz 1
Drug: Placebo
  Arms: Placebo
Drug: Oltipraz 2 (120mg)
  Arms: Oltipraz 2

SUMMARY:
Dithiolethiones, a novel class of adenosine monophosphate-activated protein kinase (AMPK) activators, prevent insulin resistance through AMPK-dependent p70 ribosomal S6 kinase-1 (S6K1) inhibition. And it is well known that the modulation of S6K1 by oltipraz inhibited the development of insulin resistance and hyperglycemia through the AMPK-S6K1 pathway.Also some research reported that LXRg (a member of the nuclear hormone receptor)-mediated increases in SREBP-1c (the sterol regulatory element-binding protein-1c gene) promote the expression of lipogenic genes and enhance fatty acid synthesis and oltipraz inhibits LXRg and SREBP-c. Therefore, Oltipraz inhibits fatty acid synthesis through AMPK-S6K1 pathway and LXRg-SREBP-1c pathway in liver.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 19 under 75 years of age
* Patients with non-alcoholic fatty liver disease except for cirrhosis
* Patients who have abnormal ALT, AST
* Patients who are satisfied with laboratory test
* Patients who agree to contraception
* Patients who can keet the diet

Exclusion Criteria:

* Over 2 ratio of AST to ALT
* Type 1 diabetes mellitus (insulin-dependent diabetes mellitus) or Type 2 diabetes mellitus(not controlled)
* Disorder in liver function with an exception of non-alcoholic fatty liver
* Patients with malignant tumors
* Patients who have been taken drugs induced fatty liver within 8 weeks of participation in this study
* Patients who has been taken any medications that could affect the treatment for NAFLD within 4 weeks
* Patients who have been taken Vitamin E (≥ 800 IU/day), thiazolidinediones, orlistat within 12 weeks
* Patients who had a Bariatric surgery less than 6 month prior to the participation in the study
* Patients who are judged by investigator that participation of the study is difficult due to disease as follow;
* Any history of immune disorder
* Patients who have received treatment that may affect liver function within 1 month prior to the participation in the study
* Patient who has been administered other investigational product within 1 month prior to the participation in the study
* Patient who is not allowed to get MRS test: pacemaker, shunt and etc
* Pregnant or nursing women
* anti-HIV antibody (+)
* Patient who considered ineligible for participation in the study as Investigator's judgment

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2014-02; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
MRS(magnetic resonance spectroscopy) | 24 weeks
  To evaluate the efficacy of the Oltipraz on change in quantity of liver fat (% change) assessed by MRS from baseline to 24 weeks in patients.

SECONDARY OUTCOMES:
change in liver fat concentration | 24 weeks
change in BMI | 8, 16, 24 weeks
change in NAFLD Fibrosis score (NFS) | 24 weeks
change in ALT, AST, γ-GT | 8, 16, 24 weeks
change in Cholesterol (total, LDL, HDL, VLDL), Triglyceride (TG) | 8, 16, 24 weeks
change in HOMA-IR | 8, 16, 24 weeks
change in waist circumference | 24 weeks

OTHER OUTCOMES:
change in Adipokine, CK-18 | 8, 16, 24 weeks

CONTACTS AND LOCATIONS:
Locations (5):
- South Korea (5):
  - NHUS Ilsan Hospital, Ilsan-ro Ilsan-donggu, Goyang-si
  - Inje University Ilsan Paik Hospital, Dahwa-dong, Ilsanseo-gu, Goyang-si, Gyeonggi-do
  - Seoul National University Hospital, Daehak-ro Jongno-gu, Seoul
  - Korea University Guro hospital, Gurodong-ro, Seoul
  - Boramae Hospital, Sindaebang-dong Dongjak-gu, Seoul